CLINICAL TRIAL: NCT03270839
Title: Motion Sickness Medications and Vestibular Time Constant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Dror Tal, Head of Motion Sickness and Human Performance Laboratory, Principal Investigator, Medical Corps, Israel Defense Force
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1723-2016
Record Dates: First submitted 2017-04-02; First posted 2017-09-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Drug Reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Meclizine; Scopolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Responsive to Scopolamine (Active) (Active Comparator): Scopolamine administration - subject will take 1 tablet per os (Kwells, Hyoscine Hydrobromide 0.3mg, 1*day )
  Interventions: Drug: Kwells
- Responsive to Scopolamine (Placebo) (Placebo Comparator): Placebo administration - subject will take 1 tablet per os (Placebo Oral Tablet, no active substance in the tablet)
  Interventions: Drug: Placebo Oral Tablet
- Non-responsive to Scopolamine (Active) (Active Comparator): Scopolamine administration - subject will take 1 tablet per os (Kwells, Hyoscine Hydrobromide 0.3mg, 1*day )
  Interventions: Drug: Kwells
- Non-responsive to Scopolamine (Placebo) (Placebo Comparator): Placebo administration - subject will take 1 tablet per os (Placebo Oral Tablet, no active substance in the tablet)
  Interventions: Drug: Placebo Oral Tablet
- Responsive to Meclizine (Active) (Active Comparator): Meclizine administration - subject will take 1 tablet per os (Bonine 25Mg Chewable Tablet, Meclizine Hydrochloride 25mg, 1*day )
  Interventions: Drug: Bonine 25Mg Chewable Tablet
- Responsive to Meclizine (Placebo) (Placebo Comparator): Placebo administration - subject will take 1 tablet per os (Placebo Oral Tablet, no active substance in the tablet)
  Interventions: Drug: Placebo Oral Tablet
- Non-responsive to Meclizine (Active) (Active Comparator): Meclizine administration - subject will take 1 tablet per os (Bonine 25Mg Chewable Tablet, Meclizine Hydrochloride 25mg, 1*day )
  Interventions: Drug: Bonine 25Mg Chewable Tablet
- Non-responsive to Meclizine (Placebo) (Placebo Comparator): Placebo administration - subject will take 1 tablet per os (Placebo Oral Tablet, no active substance in the tablet)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Bonine 25Mg Chewable Tablet — Motion sickness drug
  Other Names: Meclizine
  Arms: Non-responsive to Meclizine (Active); Responsive to Meclizine (Active)
Drug: Kwells — Motion sickness drug
  Other Names: Scopolamine
  Arms: Non-responsive to Scopolamine (Active); Responsive to Scopolamine (Active)
Drug: Placebo Oral Tablet — No active substance in the tablet
  Other Names: Placebo
  Arms: Non-responsive to Meclizine (Placebo); Non-responsive to Scopolamine (Placebo); Responsive to Meclizine (Placebo); Responsive to Scopolamine (Placebo)

SUMMARY:
Sea sickness represents a major limitation on the performance of ships' crew. One of the challenges faced by the physician in the motion sickness clinic when prescribing anti-sea sickness medication is to select the appropriate drug for the patient. Difficulties arise due to high variability in the response to different drugs. In the case of sea sickness, the current procedure is to examine the drug's efficacy in each individual during real time exposure to sea conditions.

A number of studies have documented the presence of sea sickness drug receptors in the vestibular nuclei, which determine the vestibular time constant. Two clinical vestibular tests which evaluate the time constant are the Velocity Step and OKAN tests. The purpose of the proposed study is to evaluate the influence of motion sickness drugs on the vestibular time constant, as a possible bioequivalent of drug potency in the individual subject. Eighty crew members will be recruited and divided into groups responsive and non-responsive to the sea sickness drugs scopolamine and meclizine.

Subjects having a Wiker score of 7 in waves 1 meter high without drug treatment, and no improvement in symptoms after treatment will be defined as non-responsive to sea sickness drugs. Subjects having a Wiker score of 7 in waves 1 meter high without drug treatment, and a Wiker score of 4 or less after treatment, will be defined as responsive to drug therapy.

Kwells, Bonine and placebo, will be assigned to each subject in a random, double-blind fashion. Each group will perform the Velocity Step and OKAN tests before, one and two hours after drug or placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy soldiers between the ages of 18 to 40, who suffering from sea sickness
* 48 hours prior to session without any use of medications
* Soldiers who vomit in waves 1.5 meter high without drugs treatment

Exclusion Criteria:

* Anamnestic hearing Impairment
* Ear infection of any kind
* Pathological finding in an otoneurological examination, witch will be done by a trained neurophysiologist / a physician. In any case of pathological finding, patient will be advised to continue medical assesment.
* Vision pathologies the interfere with VNG test.
* Withdrawal of informed consent by the patient of any cause.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Vestibular Time Constant Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  One of the parameters measured in step velocity test [Sec]
Step Velocity Test Gain Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  One of the parameters measured in step velocity test [0-1]
Optokinetic After Nystagmus (OKAN) Gain Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  One of the parameters measured in optokinetic test [0-1]
Optokinetic After Nystagmus (OKAN) Time Constant Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  One of the parameters measured in optokinetic test [Sec]
Optokinetic After Nystagmus (OKAN) Slow Phase velocity Sum Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  One of the parameters measured in optokinetic test [Deg/Sec]
Pupil Size Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  Using pupil size chart [Mm]
Pupil Accommodation and Convergation Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  Eye test for drugs side effects.
Side Effects Questionnaire Change/differential | Baseline at the beginning of session prior to comparator (drug/placebo) receiving, 1 hour after receiving comparator and 2 hours after receiving comparator.
  Questionnaire of drugs' side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Tal, PhD, Principal Investigator — Head of Motion Sickness and Human Performance Laboratory, Principal Investigator
Locations (1):
- Israeli Navy Medical Institute, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheung BS, Howard IP, Money KE. Visually-induced sickness in normal and bilaterally labyrinthine-defective subjects. Aviat Space Environ Med. 1991 Jun;62(6):527-31. PMID 1859339
- [Background] Adamenko VM, Evangelopoulou T, Yfantopoulos J. Kirlian photography--a tool in the diagnosing of psychopathology. J Biol Photogr. 1988 Jul;56(3):85-8. No abstract available. PMID 3182575
- [Background] Golding JF, Gresty MA. Pathophysiology and treatment of motion sickness. Curr Opin Neurol. 2015 Feb;28(1):83-8. doi: 10.1097/WCO.0000000000000163. PMID 25502048
- [Background] Ishiyama A, Lopez I, Wackym PA. Molecular characterization of muscarinic receptors in the human vestibular periphery. Implications for pharmacotherapy. Am J Otol. 1997 Sep;18(5):648-54. PMID 9303164
- [Background] Phelan KD, Nakamura J, Gallagher JP. Histamine depolarizes rat medial vestibular nucleus neurons recorded intracellularly in vitro. Neurosci Lett. 1990 Feb 16;109(3):287-92. doi: 10.1016/0304-3940(90)90009-x. PMID 2139500
- [Background] Pyykko I, Schalen L, Matsuoka I. Transdermally administered scopolamine vs. dimenhydrinate. II. Effect on different types of nystagmus. Acta Otolaryngol. 1985 May-Jun;99(5-6):597-604. doi: 10.3109/00016488509182266. PMID 4024910
- [Background] Tal D, Hershkovitz D, Kaminski G, Bar R. Vestibular evoked myogenic potential threshold and seasickness susceptibility. J Vestib Res. 2006;16(6):273-8. PMID 17726280
- [Background] Bar R, Gil A, Tal D. Safety of double-dose transdermal scopolamine. Pharmacotherapy. 2009 Sep;29(9):1082-8. doi: 10.1592/phco.29.9.1082. PMID 19698013